CLINICAL TRIAL: NCT00437307
Title: Topotecan Plus Carboplatin im Vergleich Zur Standardtherapie (Paclitaxel Plus Carboplatin Oder Gemcitabin Plus Carboplatin) in Der Therapie Von Patientinnen Mit Platin-sensitivem Rezidivierten Epithelialen Ovarialkarzinom, Peritonealkarzinom Oder Tubenkarzinom
Brief Title: Hycamtin Plus Carboplatin Versus Established Regimens for the Treatment of Ovarian Cancer Relapse
Acronym: HECTOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: North Eastern German Society of Gynaecological Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3104000
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Topotecan

ARMS (2):
- 1 (Active Comparator): Topotecan: 0,75 mg/m²/d, Tage 1-3 und Carboplatin: AUC 5 (after Cockroft and Gault formula) am Tag 3 nach Topotecan, q 21d.
  Interventions: Drug: Topotecan
- 2 (No Intervention): Paclitaxel 175 mg/m2/d, day 1 and Carboplatin: AUC 5 (after Cockroft and Gault formula), day 1, q21d OR gemcitabine 1000 mg/m2/d, day 1 and 8 and Carboplatin AUC 4 (after Cockroft and Gault formula), day 1, q 21d.

INTERVENTIONS:
Drug: Topotecan — Topotecan: 0,75 mg/m²/d, day 1-3, and Carboplatin: AUC 5 (after Cockroft and Gault Formula) on day 3 after Topotecan, q 21d
  Other Names: Hycamtin
  Arms: 1

SUMMARY:
Determination of progression free survival after 12 months of FU

Determination of total survival, response and quality of life

DETAILED DESCRIPTION:
In Germany there are two established therapy regimes for platin sensitive ovarian cancer: the combination of carboplatin and paclitaxel as well as the combination of carboplatin with gemcitabine. Choice of therapy is individual due to missing randomized comparisons between the regimes. Topotecan has shown good efficacy in second-line therapy of ovarian cancer as well as a good, especially, non-hematoxic toxicity profile. Several phase II-studies have demonstrated a synergistic effect of topotecan in combination with carboplatin exhibiting good efficacy and tolerability.

It shall be tested in this randomized phase III-study if the combination of topotecan and carboplatin shows improvement of progression-free survival in comparison to the standard regimes.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years of age with platinum-sensitive recurrent ovarian cancer occurring at least six months after completion of primary standard therapy are eligible
* Patients with measurable or assessable lesions or CA-125 ≥ 2x ULN an Eastern Co-operative Oncology Group (ECOG) performance status ≤ 2
* All patients will provide written informed consent

Exclusion Criteria:

* Patients with more than two chemotherapies in their history
* Progress less than six months after completion of primary standard therapy
* Simultaneous or planned radiation
* Any known hypersensitivity to topotecan, carboplatin, paclitaxel or gemcitabine
* Patients with infection
* Patients who are pregnant or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2007-03; Primary Completion 2013-07 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
progression-free survival | after 1 year-follow-up

SECONDARY OUTCOMES:
overall survival, efficacy and tolerability of the regimes and quality of life | during study and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jalid Sehouli, Study Chair — Charité Campus Vichow Klinikum
Locations (1):
- Charité Campus Virchow Klinikum, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No